CLINICAL TRIAL: NCT04257188
Title: A Prospective, One-center Clinical Trial to Identify the Safety and Feasibility of Sutureless Pars-plana Vitrectomy Performed in Sub-tenon Anesthesia.
Brief Title: Safety and Feasibility of Sutureless Pars-plana Vitrectomy in Sub-Tenon Anesthesia
Acronym: SAFE-VISA
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Antonis Koutsonas, Dr. med. Antonis Koutsonas, RWTH Aachen University
Other Study IDs: 19-169
Record Dates: First submitted 2019-11-19; First posted 2020-02-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Vitreoretinal Diseases
Keywords: Sub-tenon Anesthesia; Vitrectomy; Sutureless vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- minimally invasive vitrectomy under subtenon anaesthesia
  Interventions: Procedure: minimally invasive vitrectomy under subtenon anaesthesia
- minimally invasive vitrectomy under general anaesthesia
  Interventions: Procedure: minimally invasive vitrectomy under subtenon anaesthesia

INTERVENTIONS:
Procedure: minimally invasive vitrectomy under subtenon anaesthesia — The safety and feasibility in terms of tolerance and pain sensation during the surgery as well as the possible perception of light and colour sensations in minimally invasive vitrectomy under sub-tenon anesthesia shall be investigated.

SUMMARY:
The aim of this prospective study is to investigate the feasibility of performing minimally invasive vitrectomy under sub-tenon anesthesia in terms of intraoperative patients' tolerance and the surgeon's confidence. In particular, the tolerance and pain sensation during the operation as well as the possible perception of light and colour sensations are to be recorded with the help of questionnaires. In addition, the surgeon's impressions regarding eye motility, chemosis and general feasibility will be evaluated.

DETAILED DESCRIPTION:
A prospective, one-center clinical trial to identify the safety and feasibility of sutureless pars-plana vitrectomy performed in sub-tenon anesthesia.

Background:

In Germany pars-plana vitrectomies are mostly performed in general anesthesia. This requires the immediate availability of a trained anesthesiology team, which is not always granted, especially in urgent eye disease (i.e. endophthalmitis, high risk retinal detachment). Furthermore, some patients are not suitable for general anesthesia due to systemic diseases (i.e. cardio-vascular diseases). There are several procedures of local ocular anesthesia (i.e. peribulbar, retrobulbar, sub-tenon anesthesia). The main advantage of sub-tenon anesthesia is the use of a blunt cannula limiting the risk of potential complications.

Purpose:

The purpose of this study is to investigate the safety of local sub-tenon anesthesia procedure for sutureless vitrectomy (anesthetic mixture: 2ml xylocaine and 2ml bupivacaine) in a prospective clinical study design.

Objectives:

Primary outcome: The evaluation of 1. sensation of pain, 2. patients' intraoperative discomfort and 3. visual sensations using the standardized questionnaires (WONG-BAKER Faces Scale, Visual Analog Scale and individual questions).

Secondary Outcome: The evaluation of 1. chemosis, 2. eye movement, 3. surgeon's general feeling of comfort during surgery (rating scale).

ELIGIBILITY:
Inclusion Criteria:

* Age over 40 years
* Presence of a clinical condition that requires surgical treatment with vitrectomy and does not necessarily require general anesthesia (retinal detachment, endophthalmitis, vitreous hemorrhage, after silicone oil surgery, vitreomacular traction, epiretinal gliosis, macular holes, subretinal bleeding, lens luxation).

  * The medical indication for vitrectomy is not linked to study participation. Not until the patient has consented to the vitrectomy (standardized information forms) potential study subjects will be approached to participate in the clinical trial.
* Willingness to participate in the clinical trial
* Understanding the objectives of the clinical trial and the study process
* Signed informed consent form

Exclusion Criteria:

* Concomitant diseases of the eye

  * State after filtering glaucoma operations
  * Distinct corneal opacities, which make the examination considerably more difficult
  * Complicated proliferative vitreoretinopathy
* Lack of understanding of the study, its objectives and study conduct
* Psychiatric diseases
* Pregnancy
* Simultaneous participation in another clinical trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is acquired from the patient collective of the eye clinic of the University Hospital Aachen and have a medical indication for vitrectomy, which is independent of study participation.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Sensation of pain | 1 Day
  1. 11-point numeric scale ranges from '0' (means "no pain") to '10' (means "worst pain imaginable"), Questionnaire
  2. Wong-Baker FACES® Scale (6 Faces, range no hurt - hurts worst), Questionnaire
Discomfort | 1 Day
  11-point numeric scale ranges from '0' (means "no discomfort") to '10' (means "worst discomfort imaginable"), Questionnaire
Visual Sensations | 1 Day
  4 questions, Likert scale ("yes", "no", "don't know/not sure"), Questionnaire
  1. perception of details during surgery (instruments, surgeon's face)
  2. perception of colors during surgery
  3. perception of lights or shadows
  4. no light perception at all during surgery

SECONDARY OUTCOMES:
Chemosis | 1 Day
  5-point numeric scale from '0' (means no chemosis) to 4 (means chemosis of all 4 eye quadrants), Questionnaire (surgeon)
Eye movement | 1 Day
  4-point numeric scale: '0' (means ptosis and no motility), '1' (mild motility), '2' (moderate motility), '3' (full motility), Questionnaire (surgeon)
Surgeon's general feeling of comfort during the surgery | 1 Day
  6-point numeric scale ranges from '1' (means best comfort conditions) to '6' (means worst comfort conditions) Questionnaire (surgeon)

CONTACTS AND LOCATIONS:
Overall Officials: Antonis Koutsonas, Dr. med., Principal Investigator — Clinic for Ophthalmology, University Hospital RWTH Aachen
Locations (1):
- Clinic for Ophthalmology, University Hospital RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lohmann T, Baumgarten S, Prinz J, Walter P, Koutsonas A. Safety and feasibility of sutureless pars-plana vitrectomy in sub-Tenon anesthesia (SAFE-VISA): a prospective study. Eur J Med Res. 2023 Oct 30;28(1):472. doi: 10.1186/s40001-023-01447-2. PMID 37899488